CLINICAL TRIAL: NCT02944695
Title: Adherence to Safety and Infection Control Guideline in Bronchoscopy Units
Brief Title: Audit of Bronchoscopy Practice in Egypt: Adherence to Safety and Infection Control Guidelines
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Prof. Dr. Aliae AR Mohamed-Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: AssiutU1
Record Dates: First submitted 2016-10-22; First posted 2016-10-26 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Infection Control
Keywords: audit; infection control; bronchoscopy unit; Egypt

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: audit — Practice adherence to guidelines

SUMMARY:
Both patient and staff safety are of major importance during the procedure of fibreoptic bronchoscopy. Patient safety depends partly on adequate disinfection of instruments and accessories used as well as careful monitoring during the procedure.

DETAILED DESCRIPTION:
Adequate facilities, manpower and training are also essential. Staff safety depends partly on adequate procedures to minimise any risks of sensitisation to agents such as glutaraldehyde. An audit well be carried out of bronchoscopy procedures in hospitals in the Egypt and the findings well be compared with published guidelines on good practice and clinical consensus

ELIGIBILITY:
Inclusion Criteria:

* Bronchoscopy Units personnel

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Bronchoscopy Units personnel: Physicians- Nurses-workers
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of adherence to guidelines on disinfection procedures and patient monitoring | 3 months

SECONDARY OUTCOMES:
self- administered questionnaire | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Aliae Mohamed-Hussein, MD, Study Chair — Professor of Pulmonology- Faculty of Medicine-Assiut University
Locations (1):
- Pulmonology Departments, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No